CLINICAL TRIAL: NCT04982484
Title: Effects of Anti-VEGF Injections (Ranibizumab, Lucentis) on Visual Acuity, Reading Speed and Retinal Thickness in Wet-AMD Patients
Brief Title: Reading Speed Improvements in Wet-AMD Patients After Ranibizumab Treatment
Acronym: PAMER
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Collaborators: University of Pecs (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-01-UPMS
Record Dates: First submitted 2021-07-20; First posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Ophthalmopathy; Wet Macular Degeneration
MeSH Terms: conditions — Eye Diseases; Wet Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
AMD (age-related macular degeneration), is the leading cause of blindness in individuals over the age of 55. There is no cure for wet-AMD but anti-VEGF treatments significantly minimize the vision loss over time. To study the correlation between anti-VEGF injection bevacizumab (Lucentis), visual acuity, macular thickness and last but not least reading speed in wet-AMD patients.

The study was conducted on 50 eyes of 50 wet-AMD patients. Subjects were monthly treated with an intra-vitreal Lucentis injection for 3 months; further injections were given when a loss of 5 or more letters of visual acuity was observed and/or when the retinal thickness in the affected macular area increased by 100 µm. In addition to a full ophthalmological examination reading speed was investigated via the Radner reading chart before and 3 months after treatment. The collected data was analyzed using paired t-tests.

DETAILED DESCRIPTION:
Age related macular degeneration also known as AMD is the most common cause of blindness in Europe, the USA and other industrialized countries. AMD appears in people above the age of 50. The origin despite intensive research and many clinical trials is not fully understood. However, it is assumed that AMD is multifactorial. It has metabolic, genetic and environmental components that play crucial roles in the development of the disease. The interaction of different etiologic risk factors in chronic changes in the macular area (choroid, Bruch's membrane, and retinal pigment epithelium) is reflected in a slowly progressive loss of vision. AMD is classified into a dry and a wet form. The dry form represents 80% of all AMDs and it only leads to blindness in 10% of the cases. Dry AMD is characterized by drusen, pigmentary changes (hypo/hyper-pigmentation and-or atrophy of the photoreceptors with the RPE and the choriocapillaries as well). A successful therapy for this form is still unknown, but studies have shown that a change in lifestyle and dietary supplements (vitamins) can slow the progression of the disease. The wet form represents 20% of AMDs, but in 80-90% of the cases patients may experience rapid and serious vision loss. The vision loss is due to the formation of abnormal blood vessels, which are leaking in the choroid because they have no barrier and cause accumulation of blood and fluid in the intraretinal and/or subretinal space and ultimately leading to an irreversible scarring stage (Kuhnt-Junius scar). Against wet-AMD, there are numerous treatment possibilities, and they are very efficient. The treatment is mainly on the basis of anti-angiogenesis, the anti-vascular endothelial growth factor drug (Anti-VEGF) comes as an intravitreal injection ranibizumab (Lucentis). With only a few articles focusing on the reading speeds as a criteria in patients with macular disorders, analyses of the evolution of the reading speed of Wet-AMD patients are needed before and after Lucentis injections with the use Radner's reading chart : The Radner reading chart is a highly standardized multilingual reading test system that was developed in 1998 for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* AMD, Age related macular degeneration (Wet-form)

Exclusion Criteria:

* Age related macular degeneration (Dry-form)
* Diabetic macular oedema
* Other related macular oedemas

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Macular oedema due to WET-AMD
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2013-06-01 (Actual); Study Completion 2013-08-01 (Actual)

PRIMARY OUTCOMES:
Reading speed day 0 | day 0
  Reading speed measurement via Radner reading chart (a highly standardized multilingual reading test system that was developed for clinical practice and research) We measured reading speed on 50 patients before and 3 months after treatment. The reading chart consists of "sentence optotypes", which are optimized reading test items, standardized by construction and statistical selection. Sentence optotypes consist of short sentences that are highly comparable in terms of number of words (14 words), word length, and position of words, lexical difficulty and syntactical complexity. Language specific characteristics were taken into account as were the number of letters and syllables per word, line, and sentence. The advantage of such sentence optotypes is that they minimize variations between test items and keep the geometric proportions constant.
Reading speed M3 | month 3
  Reading speed measurement via Radner reading chart (a highly standardized multilingual reading test system that was developed for clinical practice and research) We measured reading speed on 50 patients before and 3 months after treatment. The reading chart consists of "sentence optotypes", which are optimized reading test items, standardized by construction and statistical selection. Sentence optotypes consist of short sentences that are highly comparable in terms of number of words (14 words), word length, and position of words, lexical difficulty and syntactical complexity. Language specific characteristics were taken into account as were the number of letters and syllables per word, line, and sentence. The advantage of such sentence optotypes is that they minimize variations between test items and keep the geometric proportions constant.

SECONDARY OUTCOMES:
Visual acuity using the ETDRS chart day 0 | day 0
  ETDRS stands for the Early Treatment of Diabetic Retinopathy Study. This landmark study helped to define the standardization of eye charts and visual acuity testing, resulting in the development of these ETDRS charts. The charts use ETDRS letters, or a geometric progression in letter size from line to line, each line being of equal difficulty.
  The ETDRS chart format has been accepted by the National Eye Institute and the FDA, and is mandated for many clinical trials performed worldwide. It is accepted worldwide as today's Gold Standard for accurate visual acuity measurement. ETDRS scoring can be accomplished in a number of different ways. The most common method is when the patient starts at the top of the chart and begins to read down the chart. The patient reads down the chart until he or she reaches a row where a minimum of three letters on a line cannot be read. The patient is scored by how many letters could be correctly identified.
Visual acuity using the ETDRS chartM3 | month 3
  ETDRS stands for the Early Treatment of Diabetic Retinopathy Study. This landmark study helped to define the standardization of eye charts and visual acuity testing, resulting in the development of these ETDRS charts. The charts use ETDRS letters, or a geometric progression in letter size from line to line, each line being of equal difficulty.
  The ETDRS chart format has been accepted by the National Eye Institute and the FDA, and is mandated for many clinical trials performed worldwide. It is accepted worldwide as today's Gold Standard for accurate visual acuity measurement. ETDRS scoring can be accomplished in a number of different ways. The most common method is when the patient starts at the top of the chart and begins to read down the chart. The patient reads down the chart until he or she reaches a row where a minimum of three letters on a line cannot be read. The patient is scored by how many letters could be correctly identified.
Maculare thickness Day0 | day 0
  Optical coherence tomography (OCT) is a non-invasive imaging test that provides anteroposterior images by measuring the echo time and intensity of reflected or backscattered light from intraretinal microstructures.
  With OCT, each of the retina's distinctive layers can be seen, allowing us to map and measure their thickness.
Maculare thickness M3 | Month 3
  Optical coherence tomography (OCT) is a non-invasive imaging test that provides anteroposterior images by measuring the echo time and intensity of reflected or backscattered light from intraretinal microstructures.
  With OCT, each of the retina's distinctive layers can be seen, allowing us to map and measure their thickness.

CONTACTS AND LOCATIONS:
Overall Officials: Georges Jr Hayek, MD, Principal Investigator — CHR Metz Thionville Hopital de Mercy